CLINICAL TRIAL: NCT05771441
Title: Effect of Heat Therapies on Pain, Functional Status, Range of Motion, and Disability in Patients With Neck Pain
Brief Title: Effects of Neck Stabilization Exercise With Heat Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Yeşil (Other)
Responsible Party: Sponsor-Investigator, Hilal Yeşil, Assoc.Prof., Afyonkarahisar Health Sciences University
Organization: Afyonkarahisar Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HYSHNP
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain
Keywords: hot pack; exercise; ultrasound therapy
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — tau-Crystallins; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- neck stabilization exercise (NSE) (Active Comparator): the patients who had NSE
  Interventions: Other: neck stabilization exercise (nse)
- NSE + HOT PACK THERAPY (Active Comparator): the patients who had NSE+ hot pack
  Interventions: Other: NSE + HOT PACK THERAPY
- NSE + infrared therapy (Active Comparator): the patients who had NSE+ infrared therapy
  Interventions: Other: NSE + infrared therapy
- NSE + ultrasound therapy (Active Comparator): the patients who had NSE+ ultrasound therapy
  Interventions: Other: NSE + ultrasound therapy

INTERVENTIONS:
Other: neck stabilization exercise (nse) — neck stabilization exercise (nse)- exercise
  Arms: neck stabilization exercise (NSE)
Other: NSE + HOT PACK THERAPY — NSE + HOT PACK THERAPY- exercise plus heat therapy
  Arms: NSE + HOT PACK THERAPY
Other: NSE + infrared therapy — NSE + infrared therapy- exercise plus heat therapy
  Arms: NSE + infrared therapy
Other: NSE + ultrasound therapy — NSE + ultrasound therapy exercise plus heat therapy
  Arms: NSE + ultrasound therapy

SUMMARY:
In this study, we aimed to determine the effects of heat therapies and neck stabilization exercises on pain, disability, range of motion, and mood of NP patients.

DETAILED DESCRIPTION:
Chronic non-specific neck pain (NP) has become one of the main causes of disability in the adult population around the world.Several treatment options used like; exercise, manual therapy, electrotherapy, and hot treatments etc. In this study, we aimed to determine the effects of heat therapies and neck stabilization exercises on pain, disability, range of motion, and mood of NP patients.100 patients with NP will be included.Patients will be randomyl assigned to 4 groups and will receive a total of 3 weeks of treatment. Patients' pain levels (visual analogoue scale VAS), quality of life (short form 36), mood (Beck deppression inventory BDI), range of motion, and neck disability index were evaluated prior to treatment, at 6th and at 12th weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic neck pain

Exclusion Criteria:

* sensory deficit on neck area, servical disc pathologies, neurological deficit, malignity, secondary causes for neck pain, active inflammation, arthritis on the neck area, serious mental health problems, pregnancy, spine surgery, and having received treatment to the cervical region in the last 6 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
change from baseline VAS (visual analog scale) at 6th and 12th week | up to 12 weeks
  The patients were asked to make an assesment of their pain level between 0 and 10 scale

SECONDARY OUTCOMES:
Change from baseline quality of life (short form 36) at 6th and 12th week | up to 12 weeks
  The physical and mental health summary scores were the primary components used. Scoring is on a scale of 0 to 100 and a higher score reflects better health-related quality of life.
Change from baseline shoulder range of motion (ROM) at 6th and 12th week | up to 12 weeks
  The patients' joint range of motion will be measured with a goniometer.
Change from baseline Beck depression inventory (BDI) at 6th and 12th week | up to 12 weeks
  A total Beck score (0-63) is obtained by giving each question a score of 0-3 in the survey. 17 is considered the threshold value for the degree of depression.
Change from baseline neck disability index (NDI) at 6th and 12th week | up to 12 weeks
  Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
  The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal Yeşil, Merkez, Afyonkarahisar, Turkey (Türkiye)